CLINICAL TRIAL: NCT03699917
Title: The Impact of Intraoperative Goal-directed Fluid Therapy on Complications After Pancreaticoduodenectomy
Brief Title: Goal-directed Fluid Therapy on Complications After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #:06-12-34E
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2018-10

CONDITIONS: Pancreaticoduodenectomy; Stroke Volume Variation
Keywords: Fluid therapy; gastric emptying; pancreatic leak; pancreaticoduodenectomy; stroke volume variation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SVV < 12: Patients undergoing pancreaticoduodenectomy with an intraoperative stroke volume variation of less than 12.
- Patients with SVV > or = 12: Patients undergoing pancreaticoduodenectomy with an intraoperative stroke volume variation of greater than or equal to 12.

SUMMARY:
Optimal fluid balance is critical to minimize anastomotic edema in patients undergoing pancreaticoduodenectomy. This study examined the effects of decreased fluid administration on rates of postoperative pancreatic leak and delayed gastric emptying.

DETAILED DESCRIPTION:
Retrospective study of 10564 patients undergoing pancreaticoduodenectomy at a single institution from January, 2015 through July, 2016. Stroke volume variation (SVV) was tracked and titrated during the procedure.

All patients were seen preoperatively in the department clinic setting, and indications for pancreaticoduodenectomy were for pancreatic adenocarcinoma, neuroendocrine tumors, chronic pancreatitis, non-adeno malignancy, and other benign. benign and malignant disease.

Patients were excluded if they had any of the following during surgery: venous resection and reconstructive involving the portal venous system; estimated blood loss exceeding two liters; high dose steroid administration; use of irreversible electroporation for margin enhancement; lack of SVV equipment or inconsistent SVV recordings; use of the robotic surgical system.

Primary outcomes measures were recorded for each patient were: pancreatic leak and delayed gastric emptying. Pancreatic leak was defined according to the international study group for pancreatic fistulas: "an external fistula with a drain output of any measurable volume after postoperative day three with an amylase level greater than three times the upper limit of the normal serum value." Delayed gastric emptying was defined clinically as persistent postoperative emesis requiring nasogastric tube placement, prokinetic agents, or hospital readmission for endoscopic gastrostomy placement.

A comparative analysis of postoperative complications was performed between patients with a median SVV < 12 during the extirpative and reconstructive phases of the procedure compared with patients with an SVV > 12. The investigators chose an SVV value of greater than 12 to represent a "dry" state because previous studies have shown that this value represents decreased fluid administration.

ELIGIBILITY:
Inclusion Criteria:

• pancreatic adenocarcinoma, neuroendocrine tumors, chronic pancreatitis, non-adeno malignancy, and other benign lesion

Exclusion Criteria:

* venous resection and reconstructive involving the portal venous system
* estimated blood loss exceeding two liters
* high dose steroid administration
* use of irreversible electroporation for margin enhancement
* lack of SVV equipment or inconsistent SVV recordings
* use of the robotic surgical system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operations were performed at a high-volume center by one of four fellowship-trained hepatopancreatobiliary surgeons using an open approach. All patients underwent an open approach for pancreaticoduodenectomy.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications (Pancreatic leak and delayed gastric emptying) | 30 days postoperatively
  Number of patients with postoperative pancreatic leak and postoperative delayed gastric emptying. Stroke volume is calculated using measurements of ventricle volumes from an echocardiogram and subtracting the volume of the blood in the ventricle at the end of a beat (called end-systolic volume) from the volume of blood just prior to the beat (called end-diastolic volume).

CONTACTS AND LOCATIONS:
Overall Officials: Dionisios Vrochides, MD, Principal Investigator — dionisios.vrochides@atriumhealth.org
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No